CLINICAL TRIAL: NCT01470937
Title: Early Diabetes Intervention Program
Acronym: EDIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kieren Mather, Associate Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9705-34
Record Dates: First submitted 2011-10-27; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes acarbose alphaglucosidase prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acarbose (Experimental): acarbose 100 mg once daily
  Interventions: Drug: Acarbose
- Placebo (Placebo Comparator): Matched placebo was administered for acarbose 100 mg once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acarbose — acarbose 100 mg PO once daily
  Other Names: Precose
  Arms: Acarbose
Drug: Placebo — acarbose placebo
  Arms: Placebo

SUMMARY:
This is an evaluation of the effect of acarbose to delay worsening of fasting glucose control in early Type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A double blind, randomized, placebo-controlled clinical trial of acarbose in subjects with type 2 diabetes (an FDA-approved indication). Subjects were identified who had diabetes by glucose tolerance test criteria but non-diabetic fasting glucose concentrations. Treatment interventions were assessed for their ability to delay worsening of fasting glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose <140 mg/dL
* 75 g OGTT 2hr glucose >120 mg/dL
* BMI > 25 OR history of gestational diabetes mellitus OR family history of type 2 diabetes
* Age at least 25 years

Exclusion Criteria:

* Cancer within 5 years
* Chronic infectious disease (HIV, Hepatitis)
* CVD event within 6 months
* Uncontrolled hypertension or requiring beta blockers or thiazide diuretics for control
* elevated AST or ALT
* Serum creatinine >1.4 mg/dL (men) or >1.3 mg/dL (women)
* TG >600 mg/dL
* Known glucosidase intolerance
* Inability to comply with protocol requirements.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 1998-02; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Progression of fasting glucose >140 mg/dL | From date of randomization until the date of first documented progression or censoring, up to 5 years post randomization
  Fasting plasma glucose was measured quarterly for up to 5 years. Two consecutive measures above 140 mg/dL defined progression.

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University; Robert V Considine, PhD, Principal Investigator — Indiana University; Marian S Kirkman, MD, Study Director — Indiana University
Locations (1):
- Indiana University Hospital GCRC, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Kirkman MS, Shankar RR, Shankar S, Shen C, Brizendine E, Baron A, McGill J. Treating postprandial hyperglycemia does not appear to delay progression of early type 2 diabetes: the Early Diabetes Intervention Program. Diabetes Care. 2006 Sep;29(9):2095-101. doi: 10.2337/dc06-0061. PMID 16936159
- [Derived] Patel YR, Kirkman MS, Considine RV, Hannon TS, Mather KJ. Changes in Weight and Glucose Can Protect Against Progression in Early Diabetes Independent of Improvements in beta-Cell Function. J Clin Endocrinol Metab. 2016 Nov;101(11):4076-4084. doi: 10.1210/jc.2016-2056. Epub 2016 Aug 17. PMID 27533307
- [Derived] Hannon TS, Kirkman MS, Patel YR, Considine RV, Mather KJ. Profound defects in beta-cell function in screen-detected type 2 diabetes are not improved with glucose-lowering treatment in the Early Diabetes Intervention Program (EDIP). Diabetes Metab Res Rev. 2014 Nov;30(8):767-76. doi: 10.1002/dmrr.2553. PMID 24819707